CLINICAL TRIAL: NCT02715011
Title: A Phase 1, First-in-Human, Open-Label, Dose Escalation Study of JNJ-63709178, a Humanized CD123 x CD3 DuoBody in Subjects With Relapsed or Refractory AML
Brief Title: Dose Escalation Study of JNJ-63709178, a Humanized CD123 x CD3 DuoBody in Participants With Relapsed or Refractory Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108147; 63709178AML1001 (Other: Janssen Research & Development, LLC); 2016-000208-27 (EudraCT Number)
Record Dates: First submitted 2016-03-16; First posted 2016-03-22 (Estimated); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Leukemia, Myeloid, Acute; JNJ-63709178
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Escalation (Experimental): Participants will receive JNJ-63709178 in Part 1 (in different cohorts). Each subsequent cohort will receive JNJ-63709178 at an increased dose level. Ascending doses may be given initially to minimize or prevent cytokine release syndrome. Dose escalation will continue until the maximum tolerated dose is reached or all planned doses are administered.
  Interventions: Drug: JNJ-63709178
- Part 2: Dose Expansion (Experimental): Participants will receive JNJ-63709178 at the recommended Phase 2 dose(s) (RP2D) determined in dose expansion phase.
  Interventions: Drug: JNJ-63709178

INTERVENTIONS:
Drug: JNJ-63709178 — Participants will receive JNJ-63709178 in Part 1 and Part 2.

SUMMARY:
The purpose of this study is to characterize the safety and tolerability of JNJ-63709178 and identify the recommended Phase 2 dose(s) (RP2D) and schedule for JNJ-63709178 in Part 1 and to characterize the safety and tolerability of JNJ-63709178 at the RP2D(s) in Part 2.

DETAILED DESCRIPTION:
This is first-in-human (FIH) Phase 1, open-label (identity of assigned study drug will be known), multicenter, dose escalation study with dose expansion to identify the RP2D and to evaluate the safety, tolerability, and preliminary antitumor activity of JNJ-63709178 in adult participants with relapsed or refractory acute myeloid leukemia (AML) who are ineligible for or have exhausted standard therapeutic options. The study will be conducted in 2 parts: dose escalation and dose expansion. The study is divided into 3 periods: a Screening Phase (within 28 days before the first dose of study drug), a Treatment Phase (first dose of study drug until the last dose of study drug) and a Post-treatment Follow-up Phase (up to the end of study participation or end of study). Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of acute myeloid leukemia (AML) according to the World Health Organization 2008 criteria with relapsed or refractory disease and ineligible for or have exhausted standard therapeutic options
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Hematology laboratory parameters within the Protocol specified range
* Chemistry laboratory parameters within the Protocol specified range
* A woman of childbearing potential must have a negative highly sensitive serum (beta human chorionic gonadotropin [b-hCG]) or urine test prior to the first dose of study drug

Exclusion Criteria:

* Acute promyelocytic leukemia
* Active central nervous system involvement
* Prior solid organ transplantation
* Prior hematopoietic stem cell transplant within 6 months of enrollment. If the participant had an allogenic transplant there must be no apparent signs of graft versus host disease and participants must have discontinued all immunosuppressive therapies for at least 4 weeks
* Prior treatment with a CD123xCD3 bispecific agent, T cells expressing CD123 specific chimeric antigen receptor, or toxin-conjugated to CD123 antibodies; prior treatment with naked anti-CD123 monoclonal antibody is permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of participants with dose-limiting toxicity (DLT) | Up to Day 28
Part 1: Type of dose-limiting toxicity (DLT) | Up to Day 28
Part 2: Number of participants with adverse events and serious adverse events | Up to 1.5 years
Part 2: Number of participants with adverse events by severity | Up to 1.5 years

SECONDARY OUTCOMES:
Part 2: Serum concentration of JNJ-63709178 | Up to 1.5 years
Part 2: JNJ-63709178 Receptor occupancy | Up to 1.5 years
Part 2: Number of participants with depletion of CD123 expressing cells | Up to 1.5 years
Part 2: Systemic cytokine concentration | Up to 1.5 years
Part 2: Concentration of markers of T cell activation | Up to 1.5 years
Part 2: Anti- JNJ-63709178 antibodies concentration | Up to 1.5 years
Part 2: Overall response rate (ORR) | Up to 1.5 years
  ORR rate is defined as the rate of complete response (CR) plus CR with incomplete recovery (CRi) plus CR with partial hematologic recovery (CRh).
Part 2: Event-free survival (EFS) | Up to 1.5 years
  EFS is defined as time from start of treatment to the date of an event, that is, first documented treatment failure, relapse from CR, CRi, or CRh, or death due to any cause.
Part 2: Relapse-free survival (RFS) | Up to 1.5 years
  RFS is defined as time from CR, CRi, or CRh confirmed objective response to relapse from CR, CRi, or CRh or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (10):
- United States (7):
  - Detroit, Michigan
  - New York, New York
  - Charlotte, North Carolina
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Nashville, Tennessee
  - Houston, Texas
- Spain (3):
  - Barcelona
  - Madrid
  - Seville